CLINICAL TRIAL: NCT02423941
Title: A Randomized Clinical Study of Retrograde Caval or Antegrade Portal Reperfusion for Early Graft Dysfunction Prevention in Deceased Brain Dead Donor Liver Transplantation
Brief Title: A Study of Retrograde rEperfusion in Dbd Donor LIver Transplantation
Acronym: REDLIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Republican Scientific and Practical Center for Organ and Tissue Transplantation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 616.36-089.843-008.6-07-037
Record Dates: First submitted 2015-04-19; First posted 2015-04-22 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Liver Transplantation; Reperfusion; Delayed Graft Function
Keywords: Liver Transplantation; Retrograde Reperfusion; Graft dysfunction; Randomized study
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retrograde reperfusion (Experimental): During the transplant procedure the liver is initially reperfused retrogradely via hepatic veins. Venting of 300 ml blood is allowed via donor portal vein. After completion the portal vein anastomosis and retrograde venting of another 100 ml blood the antegrade portal reperfusion is performed.
  Interventions: Procedure: Retrogade reperfusion
- Antegrade reperfusion (Active Comparator): During the transplant procedure the liver is reperfused conventionally, antegradely via portal vein after completion of caval and portal anastomoses. Venting of 300 ml blood is allowed via tube placed in infrahepatiс caval anastomosis before unclamping the vena cava.
  Interventions: Procedure: Antegrade reperfusion

INTERVENTIONS:
Procedure: Retrogade reperfusion — Retrogade caval reperfusion of the donor liver during the transplant procedure with consequent arterial reperfusion.
  Other Names: Caval reperfusion
  Arms: Retrograde reperfusion
Procedure: Antegrade reperfusion — Antegrade conventional portal reperfusion of the donor liver during the transplant procedure with consequent arterial reperfusion.
  Other Names: Conventional sequential portal-arterial reperfusion
  Arms: Antegrade reperfusion

SUMMARY:
To evaluate whether retrograde caval reperfusion of liver graft could be superior over antegrade portal reperfusion in regard of incidence and severity of early allograft liver dysfunction.

All eligible enrolled liver transplant candidates will be randomized to receive either:

1. retrograde caval, followed by sequential portal-arterial, reperfusion or
2. antegrade, sequential portal-arterial reperfusion.

DETAILED DESCRIPTION:
We hypothesize that retrograde caval reperfusion could be superior over antegrade portal reperfusion in regard of incidence and severity of early allograft liver dysfunction.

Chi-square method of sample size estimation with a=0,05, b=0,20 and P1-P2 = 0,25 required a 41 subject per group (Stephen B Hulley, Steven R Cummings, Warren S Browner, Deborah G Grady, Thomas B Newman.-4th ed. Lippincott Williams & Wilkins, 2013).

After signing the informed consent 90 patients will be randomized to study and active-control group (45 each).

Only patients undergoing classical technique (retrohepatic IVC resection) of liver transplantation without vena-venous bypass will be enrolled to the study.

In the study group after completion of both caval anastomoses (super and infra-hepatic) the infra-hepatic cava-clamp is released and removed allowing the filling and flushing the liver retrogradely through the hepatic veins. 300 ml of blood is drained via donor portal vein and the vein will be clamped.

Suprahepatic cava-clamp is released and removed allowing venous return to the right atrium.

Portal vein anastomosis will be constructed. Before the last 2-3 stitches another 100 ml will be drained retrogradely. Recipient portal vein clamp is removed and liver will be reperfused antegradely. After that arterial and biliary anastomoses will be constructed.

In the control group cava-clamps are not removed until completion the portal vein anastomosis.

Chi-square test and regression analysis will be used to test the difference in incidence of early allograft liver dysfunction in the study groups.

Mann-Whitney test will be used to compare the median of highest aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels 24 and 48 hours post-reperfusion.

ELIGIBILITY:
Donor Inclusion Criteria:

* deceased brain dead
* age 18-59
* length of ICU treatment up to 7 days
* highest AST and ALT up to 200 UI/L
* macroscopic steatosis up to 30%
* highest serum sodium up to 165 mmol/L
* highest bilirubin 25 µmol/L
* application of norepinephrine is allowed
* preservation solution - HTK (Custodiol)

Recipient inclusion Criteria:

* age 18-69
* primary liver transplant
* full-size transplant

Technique of liver transplant:

* with IVC resection;
* without veno-venous bypass;
* sequential portal-arterial reperfusion
* flushing of portal vascular bed with 500 ml of called to 2-4 °C saline at back-table before implantataion

Recipient exclusion Criteria:

* live donor liver transplant
* reduced and split grafts;
* multi organ failure (including fulminant and UNOS status 1);
* fulminant hepatic failure

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-01 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of early graft dysfunction (EAD) | 1-7 postoperative days
  EAD will be assessed according to Olthoff KM, et al. Liver Transpl. 2010. Severe EAD will be assessed according to P.R. Salvalaggio, et al. Transplantation Proceedings, 2012.

SECONDARY OUTCOMES:
Median aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels | 24 and 48 hours post reperfusion
Incidence of biliary strictures (anastomotic and nonanastomotic) | 90 days after liver transplant procedure
  All biliary strictures would be diagnosed by cholangiography, either ERCP or MRCP. Ulrtrasound will be used as a screening tool to assign a cholestatic patient to cholangiography.
Incidence of in-hospital mortality | 90 days after liver transplant procedure

CONTACTS AND LOCATIONS:
Overall Officials: Oleg O Rummo, MD PhD, Study Chair — RSPC for organ and tissue transplantation, Minsk 9th clinic
Locations (1):
- RSPC for organ and tissue transplantation, Minsk 9th clinic, Minsk, Belarus

REFERENCES:
- [Background] Olthoff KM, Kulik L, Samstein B, Kaminski M, Abecassis M, Emond J, Shaked A, Christie JD. Validation of a current definition of early allograft dysfunction in liver transplant recipients and analysis of risk factors. Liver Transpl. 2010 Aug;16(8):943-9. doi: 10.1002/lt.22091. PMID 20677285
- [Background] Salvalaggio P, Afonso RC, Felga G, Ferraz-Neto BH. A proposal to grade the severity of early allograft dysfunction after liver transplantation. Einstein (Sao Paulo). 2013 Jan-Mar;11(1):23-31. doi: 10.1590/s1679-45082013000100006. PMID 23579740
- [Background] Designing Clinical Research/Stephen B Hulley, Steven R Cummings, Warren S Browner, Deborah G Grady, Thomas B Newman.-4th ed. Lippincott Williams & Wilkins, 2013.-367p.]